CLINICAL TRIAL: NCT04683224
Title: A Phase 2/3 Randomized, Multicenter, Double-Blind, Placebo Controlled, Dose-Response Study to Evaluate the Safety, Immunogenicity, and Efficacy of UB-612 Vaccine in Adults
Brief Title: A Study to Evaluate the Safety, Immunogenicity, and Efficacy of UB-612 COVID-19 Vaccine
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study was withdrawn due to redesign of the protocol.
Sponsor: Vaxxinity, Inc. (Industry)
Collaborators: Diagnósticos da América S/A (DASA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UB-612-301
Record Dates: First submitted 2020-12-10; First posted 2020-12-24 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Covid-19; SARS-CoV-2; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — UB-612 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Placebo Stratum 1: 18 to 59 age group without comorbidities (Placebo Comparator): Placebo by intramuscular injection at Day 1 and 29
  Interventions: Other: Placebo
- UB-612 Stratum 1: 18 to 59 age group without comorbidities (Experimental): UB-612 by intramuscular injection at Day 1 and 29
  Interventions: Biological: UB-612
- Placebo Stratum 2: ≥60 age group without comorbidities (Placebo Comparator): Placebo by intramuscular injection at Day 1 and 29
  Interventions: Other: Placebo
- UB-612 Stratum 2: ≥60 age group without comorbidities (Experimental): UB-612 by intramuscular injection at Day 1 and 29
  Interventions: Biological: UB-612
- Placebo Stratum 3: 18 to 59 age group with comorbidities (Placebo Comparator): Placebo by intramuscular injection at Day 1 and 29
  Interventions: Other: Placebo
- UB-612 Stratum 3: 18 to 59 age group with comorbidities (Experimental): UB-612 by intramuscular injection at Day 1 and 29
  Interventions: Biological: UB-612
- Placebo Stratum 4: ≥60 age group with comorbidities (Placebo Comparator): Placebo by intramuscular injection at Day 1 and 29
  Interventions: Other: Placebo
- UB-612 Stratum 4: ≥60 age group with comorbidities (Experimental): UB-612 by intramuscular injection at Day 1 and 29
  Interventions: Biological: UB-612

INTERVENTIONS:
Biological: UB-612 — 100 µg [microgram] of an experimental study vaccine
  Arms: UB-612 Stratum 1: 18 to 59 age group without comorbidities; UB-612 Stratum 2: ≥60 age group without comorbidities; UB-612 Stratum 3: 18 to 59 age group with comorbidities; UB-612 Stratum 4: ≥60 age group with comorbidities
Other: Placebo — Placebo is a 0.9% sodium chloride (normal saline) injection
  Arms: Placebo Stratum 1: 18 to 59 age group without comorbidities; Placebo Stratum 2: ≥60 age group without comorbidities; Placebo Stratum 3: 18 to 59 age group with comorbidities; Placebo Stratum 4: ≥60 age group with comorbidities

SUMMARY:
This is a Phase 2/3, randomized, multicenter, double-blind, dose-response study to evaluate the safety, immunogenicity, and efficacy of UB 612 in 2 age groups, adults 18 to 59 and ≥60 years of age with or without comorbidities.

DETAILED DESCRIPTION:
This Phase 2/3 trial will enroll a total of 7320 male and female subjects randomized in a double-blind manner to receive either UB-612 or placebo. Assignment will be stratified by age (18 to 59 years and ≥60 years) and by presence/absence of comorbidities.

All subjects will receive 2 doses of the study vaccine, separated by 28 days, as an intramuscular (IM) injection.

Phase 2 and Phase 3 will start simultaneously; Phase 2 will enroll all Strata #1 to #4; Phase 3 will enroll Stratum #1 until the Data and Safety Monitoring Board (DSMB) has reviewed Phase 2 data through Day 43 and endorsed enrolment of Strata #2 to #4. All subjects in Phase 2 and Phase 3 will be followed for safety and efficacy.

This Phase 2/3 study also contains a Safety and Immunogenicity Cohort (N=1300) consisting of 1000 SARS-CoV-2 seronegative subjects (320 subjects enrolled in Phase 2 and 680 subjects enrolled in Phase 3) and 300 SARS-CoV-2 seropositive subjects enrolled in Phase 3.

ELIGIBILITY:
Inclusion Criteria:

1. Understands and agrees to comply with the study procedures and provides written informed consent.
2. Passes written comprehension test outlining study procedures.
3. Male or female, aged 18 to 59 years or aged >60 years at randomization.
4. Canadian Frailty Scale score of 0 to 6 (see Appendix 1).
5. Women of childbearing potential (WOCBP) and men must agree to practice medically effective contraception from 28 days before the first vaccination until 1 month after the last vaccination (i.e., a 3-month period). The acceptable effective contraception methods include the following:

   1. Barrier method (such as condoms, diaphragm, or cervical cap) used in conjunction with spermicide
   2. Intrauterine device
   3. Prescription hormonal contraceptive taken or administered via oral (pill), transdermal (patch), subdermal, or IM route
   4. Sterilization of a female participant's monogamous male partner prior to entry into the study
   5. Abstinence
6. For WOCBP, serum pregnancy test must be negative at screening; urine pregnancy test must be negative within 24 hours before vaccination.
7. Lactating female participants must agree not to breastfeed or store breast milk for 3 days after each vaccination. A substituted formula is recommended during these periods.
8. Negative serum antibodies (IgG) against SARS-CoV-2 N protein at screening except for 300 subjects in the seropositive cohort (Phase 3 only).
9. Negative result for RT-PCR screening of saliva or nasal mid-turbinate sample for SARS-CoV-2 within 2 days before vaccination.
10. At high risk of SARS-CoV-2 exposure due to occupation (e.g., health care providers, first responders, service industry workers, etc.), residence (multi-generational home, long-term care facilities, etc.), or environment with high incidence (e.g., public transportation), including geographic area.
11. Judged to be healthy or stable with pre-existing medical condition that did not require significant change in medication or hospitalization in 3 months before enrollment or who, in the judgement of the investigator are unlikely to require a significant change in therapy or hospitalization for worsening disease in the 3 months after enrollment.
12. Must be able to read, understand, and complete questionnaires in the electronic clinical outcome assessment (eCOA) system.
13. Plans to reside within study area for the duration of the study.
14. Able to comply with study procedures, in the opinion of the investigator.

Exclusion Criteria:

1. Positive for SARS-CoV-2 shedding or self-reported history of prior infection with SARS CoV-2.
2. Seropositive for SARS-CoV-2, except for 300 subjects in the seropositive cohort in Phase 3 only.
3. Moderate or severe illness and/or fever >100.4°F/38°C within 1 week before vaccination. Screening and/or study vaccination may be rescheduled at the discretion of the investigator.
4. Canadian Frailty Scale score of ≥7 (see Appendix 1).
5. History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions.
6. Coronavirus vaccines: Previous receipt of SARS-CoV-2 vaccine or other investigational coronavirus vaccine (SARS-CoV, MERS-CoV) at any time.
7. Investigational non-coronavirus vaccines: Previous receipt of an investigational vaccine (non-coronavirus) within 1 year before the planned administration of the first dose of study vaccine.
8. Licensed vaccines: Participant received or plans to receive: (a) licensed live attenuated vaccines or licensed adjuvanted (non-aluminum compound) vaccine within 28 days before or after planned administration of study vaccine, and (b) other licensed (not noted above) vaccines within 14 days before or after planned administration of study vaccine.
9. Immunosuppressive or immunodeficient state, autoimmune diseases, chronic kidney disease (with dialysis), asplenia, recurrent severe infections.
10. Individuals who receive treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, e.g., for cancer or an autoimmune disease, or planned receipt throughout the study.
11. Has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to screening (for corticosteroids ≥20 mg/day of prednisone equivalent).
12. Has received systemic immunoglobulins or blood products within 3 months prior to the day of screening.
13. Has donated ≥450 mL of blood products within 28 days prior to screening.
14. Participant received an investigational drug (including investigational drugs for prophylaxis of COVID-19) or used an invasive investigational medical device within 30 days. However, participants who received specific anti-SARS-CoV-2 monoclonal antibody products (e.g., REGN-COV2) at any time are permanently excluded, even if such product was given as part of a normal volunteer study.
15. Currently enrolled or plans to participate in another investigational study (drug, vaccine, or device) during this study.
16. Pregnant.
17. Lactating women who are unwilling or unable to withhold breastfeeding and storing milk for 3 days after each vaccination.
18. Bleeding disorder considered a contraindication to intramuscular injection or phlebotomy.
19. Tattoos or scars at the deltoid sites of IM injection that would obscure injection site reactions.
20. Behavioral, cognitive, or psychiatric disease that, in the opinion of the Principal Investigator or his or her representative physician, affects the participant's ability to understand and cooperate with all study protocol requirements.
21. Any alcohol or drug abuse over the 12 months prior to enrollment in the study that has caused medical, professional or family problems, indicated by clinical history.
22. Any other condition that, in the opinion of the Principal Investigator or his/her representative physician, could put the safety/rights of potential participants at risk or prevent them from complying with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2023-03-22 (Estimated); Study Completion 2023-03-22 (Estimated)

PRIMARY OUTCOMES:
The incidence of local reactions, solicited systemic events, AEs, MAAEs, SAEs and AESIs | Day 1 to 24 months
  Safety and Tolerability
Change in safety chemistry blood lab values for assessment of risk in Phase 3 | Phase 2 -Day 1 to Day 36
  Percentage of subjects with changes in lab values at different time points
Change in safety hematology blood lab values for assessment of risk in Phase 3 | Phase 2 -Day 1 to Day 36
  Percentage of subjects with changes in lab values at different time points
Prevention of SARS-CoV-2 infection in adults | Day 29 to 24 Month
  SARS-CoV-2 incidence based on qPCR nasopharyngeal swab
Change after second dose through the end of study in antibody titers | Month 1, 6, 12 and 24 following Dose 2
  Immunogenicity of UB-612 vaccine

SECONDARY OUTCOMES:
Prevention of COVID-19 in adults | Day 42 to 24 Month
  COVID-19 incidence confirmed by qPCR nasopharyngeal swab
Reduction in severity of COVID-19 in adults | Day 42 to 24 Month
  Efficacy of UB-612 vaccine
Prevention of COVID-19 death in adults | Day 42 to 24 Month
  Efficacy of UB-612 vaccine
Change in SARS CoV-2 shedding | Day 42 to 24 Month
  Measured by comparing the SARS-CoV-2 shedding in vaccine and placebo subjects
Immunogenicity of UB-612 vaccine in young and older adults, with or without comorbidities, and no serological or virological evidence of past infection with SARS-CoV-2 | baseline, 7 days, 6, 12, and 24 months after Dose 2
  Number of cytokine secreting spots

OTHER OUTCOMES:
Change in SARS CoV-2 infection | Month 1, 6, 12 and 24 following Dose 2
  Efficacy of UB-612 vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Gray Heppner, Study Chair — Chief Medical Officer

IPD SHARING:
Plan to Share IPD: No